CLINICAL TRIAL: NCT07111260
Title: Comparison of the Efficacy of Hemoadsorption Combined With Hemodialysis of Different Treatment Durations in Clearing Protein-Bound Uremic Toxins: A Randomized Crossover Controlled Trial
Brief Title: Efficacy of pHA130 Hemoadsorption for 4 Hours (p4H Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Li Zuo, Director, Peking University People's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025PHB095-001
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Hemoadsorption; Duration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-Hour HA Group (Experimental): Subjects receive high-flux hemodialysis (HFHD) twice a week and hemoadsorption combined with HFHD (HAHD) once a week. The HAHD session, using a pHA130 cartridge, lasts for the entire 4-hour duration of the dialysis session. Blood flow rate is maintained at 250-350 mL/min, consistent with the patient's original HD prescription.
  Interventions: Device: pHA130 Hemoadsorption + High-Flux Hemodialysis
- 2-Hour HA Group (Active Comparator): Subjects receive high-flux hemodialysis (HFHD) twice a week and HAHD once a week. The hemoadsorption component, using a pHA130 cartridge, is performed for the first 2 hours of the session, after which the pHA130 cartridge is removed and the patient continues with standard HFHD for the remaining 2 hours. Blood flow rate during HA is 200-250 mL/min.
  Interventions: Device: pHA130 Hemoadsorption + High-Flux Hemodialysis

INTERVENTIONS:
Device: pHA130 Hemoadsorption + High-Flux Hemodialysis — A combination blood-purification procedure in which a pHA130 hemoperfusion cartridge is connected in series with a high-flux hemodialyzer. Blood first passes through the HP cartridge to adsorb protein-bound uremic toxins and is then dialyzed. In the 4-hour arm the HP cartridge remains online for the entire 4-hour session; in the 2-hour arm the cartridge is removed after 2 hours and dialysis continues alone for the remaining 2 hours. Blood-flow rates are 250-350 mL/min (4-hour arm) or 200-250 mL/min (2-hour arm).

SUMMARY:
This is an open-label, randomized, crossover study to evaluate the efficacy of extending the duration of hemoadsorption (HA) combined with hemodialysis (HD) from 2 hours to 4 hours for clearing protein-bound uremic toxins, such as Indoxyl Sulfate (IS), in stable maintenance hemodialysis patients. Patients will be randomized to receive either 2-hour HA or 4-hour HA once a week for 8 weeks, then cross over to the other treatment for another 8 weeks after a 2-week washout period. The primary endpoint is the reduction rate of IS.

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD) on maintenance hemodialysis (MHD) have a high burden of uremic toxins, particularly protein-bound uremic toxins (PBUTs), which are poorly cleared by conventional dialysis and are associated with high cardiovascular mortality. hemoadsorption (HA) is an adjunctive blood purification technique effective at removing PBUTs. The standard duration for HA sessions is typically 2-2.5 hours. However, emerging evidence suggests that extending the treatment duration may enhance toxin removal. This study aims to rigorously compare the efficacy and safety of a 4-hour HA session combined with hemodialysis against a standard 2-hour session in clearing key PBUTs like Indoxyl Sulfate (IS) and p-Cresyl Sulfate (PCS). The findings will provide crucial evidence for optimizing HA treatment protocols to improve toxin clearance and potentially patient outcomes in the ESRD population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years, regardless of gender
* Stable maintenance hemodialysis for ≥3 months, with a relatively fixed dialysis regimen
* Receiving hemodialysis 3 times per week, each session lasting ≥4 hours
* Single-pool Kt/V (spKt/V) ≥1.2 within 8 weeks prior to enrollment
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Life expectancy less than 1 year
* White blood cell count < 4 × 10⁹/L and/or platelet count < 60 × 10⁹/L
* Active or chronic gastrointestinal bleeding, or diagnosed coagulation disorders
* Active malignant tumor
* Active infection
* Pregnant or breastfeeding
* Participation in another clinical trial within the past month or currently enrolled in one
* Deemed unsuitable for the study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Reduction Rate of Serum Indoxyl Sulfate (IS) | At Week 1, Week 8, Week 11, and Week 18; blood samples will be collected at 0 hours (before treatment), 2 hours after treatment begins, and 4 hours (end of treatment) during each visit
  The reduction rate (RR) of serum Indoxyl Sulfate (IS) after a single HAHD treatment session. The RR is calculated as: RR(%) = (1 - (Post-treatment Concentration / Pre-treatment Concentration)) × 100. Post-treatment concentration will be corrected for hemoconcentration.

SECONDARY OUTCOMES:
Reduction Rate of p-Cresyl Sulfate (PCS) | At Week 1, Week 8, Week 11, and Week 18; blood samples will be collected at 0 hours (before treatment), 2 hours after treatment begins, and 4 hours (end of treatment) during each visit
  RR of serum PCS after a single session
Change from Baseline in Pre-dialysis IS levels | Baseline (Week 1) to end of period 1 (Week 8); Baseline of period 2 (Week 11) to end of period 2 (Week 18)
  Change in pre-dialysis serum concentrations of IS from the beginning to the end of each 8-week treatment period
Change from Baseline in Pre-dialysis PCS levels | Baseline (Week 1) to end of period 1 (Week 8); Baseline of period 2 (Week 11) to end of period 2 (Week 18)
  Change in pre-dialysis serum concentrations of PCS from the beginning to the end of each 8-week treatment period
Clearance of Other Uremic Toxins | Week 1, Week 8, Week 11, Week 18
  Reduction rates and/or clearance of urea, creatinine, β2-microglobulin, C-reactive protein (CRP), and Interleukin-6 (IL-6)
Number of Participants With Adverse Events, Circuit Coagulation, and Abnormal Changes in Vital Signs or Laboratory Parameters | Throughout the entire study duration (up to 18 weeks)
  All adverse events (AEs) reported during the study will be recorded and assessed for severity and relationship to the intervention. Specific safety indicators include the incidence of circuit coagulation, decreases in white blood cell count, platelet count, and hemoglobin levels, as well as changes in vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, Principal Investigator — Renal Division, Department of Medicine, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No